CLINICAL TRIAL: NCT05804656
Title: A Randomized, Double-blind, Active-controlled, Multi-center Phase 3 Trial to Investigate the Efficacy and Safety of CKDB-501A in Subjects With Moderate-to-severe Glabellar Lines
Brief Title: Efficacy and Safety of CKDB-501A in Subjects With Moderate-to-severe Glabellar Lines in Phase 3 Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CKD Bio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKDB-BAGL-301
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKDB-501A (Experimental)
  Interventions: Drug: CKDB-501A
- Botox® (Active Comparator)
  Interventions: Drug: Botox®

INTERVENTIONS:
Drug: CKDB-501A — Intramuscular injection CKDB-501A
  Arms: CKDB-501A
Drug: Botox® — Intramuscular injection Botox®
  Arms: Botox®

SUMMARY:
A Randomized, Double-blind, Active-controlled, Multi-center Phase 3 Trial to Investigate the Efficacy and Safety of CKDB-501A in Subjects with Moderated-to-severe Glabella Lines

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with at least moderate glabellar lines at maximum frown as determined by severity score of at least 2-point (moderate) on the Facial Wrinkle Scale (4-point FWS) as assessed by investigator.

Exclusion Criteria:

1. Any medical condition that can affect the neuromuscular function
2. History of facial nerve paralysis or ptosis
3. Significant facial asymmetry
4. Subjects whose glabellar lines cannot be sufficiently improved by physical method
5. Subjects who have a previous surgical history that could result in any anatomical changes related to corrugator muscle, procerus muscle, or any relevant nerves
6. Subjects with skin abnormalities at potential injection sites

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a ≥ 2-point improvement on the FWS score at maximum frown from baseline, as assessed by the investigator post-administration of the investigational product | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Beomjoon Kim, Principal Investigator — Chung-Ang University Hosptial
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi SY, Kim BJ, Lee YW, Kim WS, Yoon YN, Kim JS. Efficacy and Safety of CKDB-501A in Treating Moderate-To-Severe Glabellar Lines: A Randomized, Double-Blind, Active-Controlled, Multi-Center Phase III Trial. J Cosmet Dermatol. 2025 Jul;24(7):e70305. doi: 10.1111/jocd.70305. PMID 40586136